CLINICAL TRIAL: NCT04729465
Title: The Effect of BIS-guided Propofol Induction on the Peroperative and Postoperative Hemodynamic Response in Patients With Cardiac Risk in Ear-nose-throat Surgery.
Brief Title: The Effect of BIS-guided Propofol Induction on Hemodynamic Response in Patients With Cardiac Risk.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Fatih Yılmazer, Department of Anesthesiology, Resident, MD., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10/01/2020-5208
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia, General
Keywords: BIS, propofol, anesthesia
MeSH Terms: interventions — Propofol; Consciousness Monitors

STUDY DESIGN:
Intervention Model Description: Drug: Propofol Device : Bispectral Index Monitor
Who Masked: Participant
Masking Description: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Active Comparator: Control Patients with cardiac disaese receive general anesthesia with Propofol
  Interventions:
  Drug: Propofol
  Interventions: Drug: Propofol
- Experimental (Experimental): Experimental: Bispectral Index Monitor Patients with cardiac disease receive a general anesthesia with Propofol where the amount of anesthetics administered is decided taking into consideration the Bispectral Index Monitor.
  Interventions:
  Drug: Propofol Device: Bispectral Index Monitor
  Interventions: Drug: Propofol; Device: Bispectral Index Monitor

INTERVENTIONS:
Drug: Propofol — Propofol
Device: Bispectral Index Monitor — Bispectral Index Monitor
  Arms: Experimental

SUMMARY:
Anesthesia induction will be started by monitoring ECG, non-invasive artery monitoring, peripheral oxygen saturation and BIS for all patients who are taken to the operating room without sedation. The patients were divided into 2 groups: Group P; Propofol 2 mg / kg bolus (in 10 seconds), Group B; Propofol will be started as an infusion dose of 0,25 mg / kg / min and will be discontinued when the BIS reaches a minimum value of 60. Noninvasive arterial blood pressure and heart rate will be measured at 2-minute intervals during the first 10 minutes of induction and then at 15th , 20th ,30th and 60th minutes peroperatively. Hypotension; mean arterial pressure (MAP) <60 mmHg, bradycardia heart rate <60 / min, hypertension MAP> 120 mmHg and tachycardia heart rate> 100 / min were defined. The difference of changes, their duration, the difference between the maximal value and the baseline value, and the number of occurrences of hypotension, hypertension, and arrhythmias during the entire induction and perioperative period will be recorded. Noninvasive arterial blood pressure and heart rate measurements of the patients will be made in the postoperative period at 5th , 15th , 30th minutes and at 1st , 2nd , 4th , and 24th hours. At the end of the 1st month, it will be questioned whether the patients encounter a cardiovascular problem that will require treatment or hospitalization in the period following the surgery. All patients will be started with 5 ml / kg / hour IV crystalloid infusion. When the MAP falls below 60 mmHg during induction, the patient will be given the Trendelenburg position and the crystalloid infusion will be increased to 10 ml / kg / hour, and vasoconstrictor drug will be added if the hypotension does not improve within the following 10 minutes.

DETAILED DESCRIPTION:
surgeries performed on patients participating in the study

minor elective ear nose throat surgery (microlaryngeal surgery, biyopsy for ENT malignancy, myringoplasty)

exclusion criteria;history of stroke, stupor, dementia, long-term use of central nervous system (CNS) activator drugs, benzodiazepines and/or opiates therapy, and pregnant females

ELIGIBILITY:
Inclusion Criteria:

The patients with a cardiovascular problem requiring ENT surgery lasting less than 2 hours

Exclusion Criteria:

Patients having history of stroke, stupor, dementia, long-term use of central nervous system (CNS) activator drugs, benzodiazepines and/or opiates therapy, and pregnant females were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-08 (Estimated); Primary Completion 2021-07-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Propofol consumption | 30 minutes-2 hours
  amount of Propofol consumption during the induction of anesthesia and perioperative period with or without BIS monitoring

SECONDARY OUTCOMES:
Hemodynamic alterations | 30 minutes- 2 hours
  to observe hemodynamic alterations during propofol induction with or without BIS monitoring .